CLINICAL TRIAL: NCT00481286
Title: Improving Outcomes for Multiple Morbidities Using Collaborative Group Clinics to Empower Older Patients
Brief Title: Improving Outcomes Using Collaborative Group Clinics to Empower Older Patients
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); M.D. Anderson Cancer Center (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aanand Naik, Associate Professor, Medicine-Health Srvcs Research, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20437; 7U18HS016093 (AHRQ)
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2009-10

CONDITIONS: Diabetes; Hypertension
Keywords: Group clinics; Goal setting; Diabetes; Hypertension; Age 50+
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Clinic (Experimental): Patients in Group Clinic arm will meet every 3rd week for 12 weeks, for a total of 4 visits. At each visit, BP will be measured, home BP and glucose measurements collected. Each visit will include group-based education and feedback sessions, with an individualized process of selecting and modifying process of care goals for systolic BP, H1C, and LDL cholesterol. Short-term health behavior change goals will also be discussed.
  Interventions: Behavioral: Improving outcomes using group clinics for older patients
- Uusual Care (Placebo Comparator): Older diabetes patients will attend regular clinician visits and one targeted primary care physician visit during the 12 weeks post-enrollment. They will be enrolled in a diabetes education class. Blood pressure, H1C and lipids will be measured at enrollment, 6 weeks , and 12 weeks.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Improving outcomes using group clinics for older patients — Collaborative group clinics to empower older patients to adopt goal-setting behaviors with their health care providers and improve their diabetes-related outcomes.
  Other Names: Diabetes Group Clinic; Goal-setting Clinic
  Arms: Group Clinic
Behavioral: Standard of Care — Standard of care for diabetes patients
  Other Names: Diabetes usual care
  Arms: Uusual Care

SUMMARY:
The purpose of this study is to determine if group clinics help older veterans change behaviors with the goal of improving diabetes outcomes.

DETAILED DESCRIPTION:
Among persons aged 55-84 years, over 65% have one to three common medical conditions (e.g., hypertension, diabetes, arthritis, stroke, heart disease, etc.). Fortunately, large randomized clinical trials have demonstrated the effectiveness of treatment and prevention strategies for many chronic conditions (e.g., dietary modification and medications for hypertension, intensive glucose monitoring with diet and medication regimens for diabetes, etc.). Despite the significant findings from numerous clinical trials, most older persons continue to suffer from uncontrolled hypertension, hyperglycemia, and other predictors of poor health outcomes. Non-compliance with clinical guidelines by providers (i.e. clinical inertia) and non-adherence to doctors' recommendations are typically blamed for these unacceptably poor outcomes. For older adults with several conditions, the processes of patient-clinician collaboration are not well understood. Goal-setting behaviors may improve health care by linking desired outcomes (i.e., reduce risk of heart attacks) to the goals of care (i.e., salt restriction for hypertension control). Furthermore, the process of goal-setting may be more effective if patients internalize the importance of a particular goal and prioritize that goal among multiple clinical problems (i.e., hypertension care for patients with diabetes.

Effective methods of implementing collaborative goals and training patients to negotiate shared goals and goal-directed behaviors with their clinicians have been developed for diabetes control. The effectiveness of these methods may be enhanced through the use of clinics that enroll small groups of subjects with rapid follow-up for several weeks. Group clinics have demonstrated improved outcomes for common chronic conditions. Evidence demonstrating the synergistic benefit of efficient group clinics and collaborative goal-setting is limited. However, an approach combining these methodologies may provide an improved method of rapidly controlling multiple chronic conditions and maintaining control of those chronic conditions over a prolonged time period.

To address the gap in the implementation of effective and efficient medical care, we will develop and test a model of collaborative group clinics that empowers older patients to adopt goal-setting behaviors, increases communication with their health care provider, and improves their diabetes-related outcomes. The objectives are to use a collaborative group clinic to: 1) Improve diabetes process of care outcomes over a 3 month time period; 2) Significantly improve the maintenance of diabetes process of care improvements over a 12 month time period; and 3) Significantly improve use of self-management behaviors for diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes and hypertension
* HgA1C value greater than or equal to 7.5
* Creatinine value less than or equal to 2.0mg/dl
* SBP greater than or equal to 140

Exclusion Criteria:

* Prior diagnoses of dementia using ICD-9 codes validated for a VA population

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure; change in Hemoglobin A1C; change in low density lipoprotein | 12 months
  Change in systolic blood pressure; change in Hemoglobin A1C; change in low

SECONDARY OUTCOMES:
Attainment of benchmark levels for SBP, A1C, LDL; self-management performance (self-report); completion of group clinic | 12 months
  Attainment of benchmark levels for SBP, A1C, LDL; self-management

CONTACTS AND LOCATIONS:
Overall Officials: Aanand D Naik, MD, Principal Investigator — Baylor College of Medicine

REFERENCES:
- [Derived] Teal CR, Haidet P, Balasubramanyam AS, Rodriguez E, Naik AD. Measuring the quality of patients' goals and action plans: development and validation of a novel tool. BMC Med Inform Decis Mak. 2012 Dec 27;12:152. doi: 10.1186/1472-6947-12-152. PMID 23270422
- [Derived] Naik AD, Palmer N, Petersen NJ, Street RL Jr, Rao R, Suarez-Almazor M, Haidet P. Comparative effectiveness of goal setting in diabetes mellitus group clinics: randomized clinical trial. Arch Intern Med. 2011 Mar 14;171(5):453-9. doi: 10.1001/archinternmed.2011.70. PMID 21403042